CLINICAL TRIAL: NCT00947713
Title: Comparison of Micro-dose Human Chorionic Gonadotropin (hCG) With HMG in PCOs Patients With Previous Clomiphene Citrate (CC)-Resistant Anovulation
Brief Title: Comparison of Micro-dose Human Chorionic Gonadotropin (hCG) With Human Menopausal Gonadotropin (HMG) in Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi, Chief, Royan institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Royan-Emb-002
Record Dates: First submitted 2009-07-25; First posted 2009-07-28 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2010-04

CONDITIONS: Endocrine System Diseases; Gonadal Disorders
Keywords: Human chorionic gonadotropin; Clomiphene citrate; chronic anovulation; Polycystic Ovary Syndrome; Follicolugenesis
MeSH Terms: conditions — Endocrine System Diseases; Gonadal Disorders; Polycystic Ovary Syndrome | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose hCG group (Experimental)
  Interventions: Drug: low dose human chorionic gonadotropin
- Clomiphen citrate plus HMG (Active Comparator)
  Interventions: Drug: Clomiphen citrate plus HMG

INTERVENTIONS:
Drug: low dose human chorionic gonadotropin — patients will receive low dose human chorionic gonadotropin (HCG) in combination with clomiphen citrate
  Other Names: human chorionic gonadotropin
  Arms: Low dose hCG group
Drug: Clomiphen citrate plus HMG — patients will receive Clomiphen Citrate plus HMG
  Arms: Clomiphen citrate plus HMG

SUMMARY:
The purpose of this study is to compare the effectiveness of low dose human chorionic gonadotropin (HCG) in combination with clomiphen citrate to induce ovulation and its endocrine response in patients who had previously failed to ovulate on clomiphen citrate alone. The investigators will also compare the effectiveness and endocrine response of this approach with the regimen of adding HMG to clomiphen citrate.

DETAILED DESCRIPTION:
Infertile women with PCOS, who have showed resistance to Clomiphen Citrate (150 mg- 5 days) in a previous IUI treatment cycle at Royan Institute (Infertility and Reproductive Medicine Research Centre) will enroll in this prospective randomized clinical trial study and will randomly be divided into three groups.

The study protocol will be assessed by an independent institutional review board and Royan ethics committee. All subjects will be given the written informed consent.

Control group (CC/hMG) will receive the 100 mg CC on days 3 to 7 of that cycle but will receive 150 mg human menopausal gonadotropin (HMG) during days of 7, 8, and 9. One of experimental Group (group B) will receive a 100 mg dose of CC but will receive a 200 IU Human chorionic gonadotropin (hCG; Choriomon; IBSA, Switzerland) intramuscular injection daily when the largest follicle is 12 mm or larger mean diameter. Other experimental group (Group C) will receive a 100 mg dose of CC but will receive a 200 IU Human chorionic gonadotropin (hCG; Choriomon; IBSA, Switzerland) intramuscular injection daily From day 9(without attention to follicle size). In both experimental groups HCG administration will be continued until the largest follicle is 18-20 mm.

Ultrasound measurements of follicle number and growth, ovulation, gestational sac, and serum hormonal levels will be recorded and compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS diagnosed by the Rotterdam criteria
* Previously documented dominant follicle or follicles (R12 mm mean diameter) on transvaginal Ultrasound follicular monitoring while receiving CC at the 150-mg dose in our clinic but have failed to ovulate;
* Primary infertility
* Documented normal uterine cavity and patent tubes by either hysterosalpingogram or laparoscopy and hysteroscopy;
* Male partner had to have a normal semen analysis by World Health Organization criteria.

Exclusion Criteria:

* previous history of IVF or ICSI treatments.
* History of hormonal treatment within recent three month (Except OCP, progesterone).
* History of ovarian cutter or Ovarian drilling.
* BMI higher than 30.
* The presence of ovarian cyst (more than 30 mm) during third cycle ultrasound.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Multiple pregnancy rates, OHSS rate | Within 20 months after recruiting

SECONDARY OUTCOMES:
Pregnancy rate | Within 20 months after recruiting
The total dose of ovarian stimulation drugs | Within 20 months after recruiting
The number of embryos available for transfer | Within 20 months after recruiting
The embryo implantation rate and The live birth rate | Within 20 months after recruiting

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Ashrafi, Principal Investigator — Royan institute, Reproductive Medicine Research Centre, ACECR
Locations (1):
- Royan institute, Reproductive Medicine Research Centre, ACECR, Tehran, Tehran Province, Iran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org